CLINICAL TRIAL: NCT06888869
Title: The Development and Verification of an Interactive Home-based Rehabilitation Exercise Assessment Platform and Exploration of Technology Acceptance and Clinical Effects in Patients with Parkinson's Disease
Brief Title: Interactive Home-based Rehabilitation Exercise Assessment Platform and Exploration of Clinical Effects in Patients with Parkinson's Disease
Acronym: PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-12-004A
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; visual feedback; Exercise intervention
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Clinical rehabilitation (Experimental): Participants in this group would be treated with exercise rehabilitation for twice a week, total 12 weeks in the hospitals.
  Interventions: Other: Other: Clinical rehabilitation group
- Active Comparator: Home-based rehabilitation (Active Comparator): Rehabilitation training for twice a week, total 12 weeks at home.
  Interventions: Other: Other: Home-based rehabilitation group
- No Intervention: Control (No Intervention): The control group received Parkinson's disease treatment-related medication and was asked to maintain daily activities according to their usual lifestyle.

INTERVENTIONS:
Other: Other: Clinical rehabilitation group — Rehabilitation training for twice a week, total 12 weeks in hospitals.
  Arms: Experimental: Clinical rehabilitation
Other: Other: Home-based rehabilitation group — Rehabilitation training for twice a week, total 12 weeks at home.
  Arms: Active Comparator: Home-based rehabilitation

SUMMARY:
This study aims to develop an "Interactive Home-based Rehabilitation Exercise Assessment Platform" that incorporates visual feedback similar to virtual reality into rehabilitation machines and aerobic cycling programs. In the clinical research part, 92 Parkinson's disease patients will be randomly assigned to three groups: the clinical rehabilitation group, the home-based rehabilitation group, and the control group. Each group will undergo the intervention twice a week, with each session lasting about 30-45 minutes over a period of 12 weeks for a total of 24 combined resistance and aerobic rehabilitation training sessions. The effectiveness evaluation will include measurements of upper limb grip strength, lower limb muscle strength, the 3-meter sit-to-stand test, the 6-minute walk test, the Parkinson's Disease Severity Scale, the Quality of Life Scale, the 10-meter walk test, and technology acceptance forms.

DETAILED DESCRIPTION:
Background and Purpose: Previous research on technological interventions in exercise therapy for Parkinson's disease has shown that incorporating visual feedback through virtual reality into rehabilitation exercise programs can improve patients' balance, muscle strength, gait, and other functional performances. This study aims to develop an "Interactive Home-based Rehabilitation Exercise Assessment Platform" that incorporates visual feedback similar to virtual reality into rehabilitation machines and aerobic cycling programs. The platform uses sensors and interactive games to guide correct rehabilitation movements. The effectiveness of the platform will be validated through engineering-related tests and clinical trials further to investigate its clinical benefits for Parkinson's disease patients.

Methods: This study consists of two parts: platform development and validation and clinical research. The platform will be implemented for use in medical institutions and at home, specifically at Taipei Veterans General Hospital, utilizing six rehabilitation machines and aerobic bicycles, as well as home-based cycling combined with resistance band training. Interactive game software and laser sensors will be developed. Sensors will collect patients' physiological parameters during the rehabilitation process to ensure safety and provide real-time feedback on movements and time control during the sessions. The collected data, including angle values, cycling revolutions, and physiological parameters, will be verified for usability using commercially available products.

In the clinical research part, 92 Parkinson's disease patients will be randomly assigned to three groups: the clinical rehabilitation group, the home-based rehabilitation group, and the control group. Each group will undergo the intervention twice a week, with each session lasting about 30-45 minutes over a period of 12 weeks for a total of 24 combined resistance and aerobic rehabilitation training sessions. The effectiveness evaluation will include measurements of upper limb grip strength, lower limb muscle strength, the 3-meter sit-to-stand test, the 6-minute walk test, the Parkinson's Disease Severity Scale, the Quality of Life Scale, the 10-meter walk test, and technology acceptance forms. Statistical analysis will be performed using one-way ANOVA and chi-square tests to analyze personal data characteristics. For clinical effectiveness analysis, a two-way (group by time) ANOVA with repeated measures will be used to examine differences between groups and over time, with Bonferroni tests for post-hoc comparisons. All data will be analyzed using SPSS version 24, with a p-value of less than 0.05, which is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with primary Parkinson's disease by a neurologist
2. Modified Hoehn and Yahr Scale I-III
3. Aged 45-85 years old
4. Mini-Mental State Examination (MMSE) score of 24 or above
5. Stable on Parkinson's disease-related medications
6. Able to walk independently or use assistive devices to walk 15 meters
7. Able to understand the movements and test items
8. Able to understand and willing to sign the informed consent form

Exclusion Criteria:

1. Rheumatic diseases
2. Unstable heart and respiratory diseases (such as angina pectoris, pulmonary embolism, etc.)
3. Severe or unstable neurological or orthopedic diseases (such as stroke, dementia, fractures, etc.)
4. Severe hearing or visual impairment, unable to cooperate with researchers
5. People diagnosed with mental illness
6. People with a history of epilepsy or a direct blood relative with a history of epilepsy
7. Pregnant or breastfeeding women
8. People with any uncontrolled chronic diseases that may cause safety concerns
9. People living without family members or case caregivers.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-03-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Timed Up and Go test (TUG) at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The time score is lower, means the gait function is better.
Change from Baseline muscle strength of upper limbs at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The muscle strength of upper limbs score is higher, means the upper limbs is better.
Change from Baseline muscle strength of lower limbs at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The muscle strength of lower limbs score is higher, means the upper limbs is better.
Change from Baseline gait Speed at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The gait Speed time score is lower, means the gait function is better.
Change from Baseline the Mini-Mental State Exam (MMSE) at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The Mini-Mental State Exam score is higher, means the Cognitive function is better.
Change from Baseline Quality of Life Scale(PDQ39) at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  Quality of Life Scale score is higher, means the Quality of Life is better.
Change from Baseline technology acceptance forms at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  Technology acceptance forms score is higher, means theTechnology acceptance is better.
Change from Baseline The unified Parkinson's disease rating scale(UPDRS) at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The unified Parkinson's disease rating scale(UPDRS) score is lower, means Disease severity is better.
Change from Baseline IPAQ Taiwan Activity Survey at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  No score in this IPAQ Taiwan Activity Survey form.
Change from Baseline Six-minute walk distance at 12 weeks | pre-test(first time) and post-test(after 12 weeks)
  The Six-minute walk distance time score is lower, means walk distance is better.

IPD SHARING:
Plan to Share IPD: No